CLINICAL TRIAL: NCT01350817
Title: Randomized Open Non Comparative Multicenter Phase II Study of Sequential Erlotinib With Docetaxel Versus Docetaxel Alone in Second Line of Treatment in Patients With Non Small Cell Lung Cancer After Failure of First Line Chemotherapy
Brief Title: Erlotinib and Docetaxel in Second Line of Treatment in Patients With Non Small Cell Lung Cancer
Acronym: TARSEQ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I10004
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Erlotinib (Experimental)
  Interventions: Drug: Erlotinib + docetaxel

INTERVENTIONS:
Drug: Erlotinib + docetaxel — docetaxel :75 mg/m² IV day 1 every 3 weeks with erlotinib:150 mg/d per os d2-d16
  Arms: Erlotinib
Drug: Docetaxel — docetaxel :75 mg/m² IV day 1 every 3 weeks.
  Arms: Docetaxel

SUMMARY:
This 2 arms study will compare the efficacy and safety of treatment with sequential erlotinib plus docetaxel therapy versus docetaxel alone as second line treatment in patients with recurrent non-small cell lung cancer. Patients will be randomized to receive in group 1(experimental arm): docetaxel :75 mg/m² IV day 1 every 3 weeks with erlotinib:150 mg/d per os d2-d16 and group 2 (control arm): docetaxel :75 mg/m² IV day 1 every 3 weeks.

The anticipated time on study treatment is until disease progression. Target sample size is 156.

The main of this study is to determine the relevance of the association sequential erlotinib and docetaxel in terms of progression-free survival .

DETAILED DESCRIPTION:
In this study, the patient will be randomized in group 1(experimental arm): docetaxel :75 mg/m² IV day 1 every 3 weeks with erlotinib:150 mg/d per os d2-d16 and group 2 (control arm): docetaxel :75 mg/m² IV day 1 every 3 weeks.

Assessment during treatment: Physical examination, ECG,: every 3 weeks, laboratory tests: weekly, every 3 weeks pulmonary X-ray .The CT scans:. Measurable targets are assessed by RECIST compared to the beginning of treatment: at 6 weeks (day 42 EVA 2), 12 weeks (D84 EVA 3), 15 weeks (D105 EVA 4: Evaluation of the SSP) and then every 6 weeks until progression.

Quality of life will be assessed Day 42 then every 6 weeks during chemotherapy, Tolerability will be assessed at each visit based on CTC v4.0 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC (
* Mutational status of EGFR : wild type or unknown
* Stage IV disease with cytologic or histologic documentation in patients with a single easily accessible metastasis or metastatic relapses in a non irradiated region from a primary tumor treated with surgery or radiotherapy (with cytologic or histologic documentation of relapse)
* Presence of at least one measurable target lesion (one dimension) in a non irradiated region (at least 10 mm on spiral computed tomography).
* Age ≥ 18 years
* Performance status 0,1,2 exception : age > 74 years only PS 0 or 1
* Normal hepatic function
* Normal renal function
* Normal calcemia
* Normal haematological function
* Life expectancy > 12 weeks.
* Women of child bearing potential must use effective contraception.
* Men might be surgically sterile or accept to use an effective contraceptive procedure during and until 6 months after the treatment.
* Written informed consent to participate in the study.

Exclusion Criteria:

* PS > 2, exception : age > 74 years only PS ≥ 2
* Presence of another cancer
* Previous treatment with an anti egfr agent or docetaxel
* QT prolongation (>470 ms)
* Uncontrolled arterial hypertension.
* Concurrent radiotherapy, except for palliative bone irradiation.
* Stroke less than 6 months before study entry.
* Psychiatric or neurological disorders preventing the patient from understanding the nature of the trial
* Uncontrolled infection.
* Caval syndrome
* Other organic disorders preventing inclusion in the trial
* Malabsorption syndrome
* Allergy to erlotinib or one of its constituents
* Allergy to docetaxel or one of its constituents
* Pregnancy and breast-feeding
* Surgery less than two months before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 15 weeks. | at 15 weeks

SECONDARY OUTCOMES:
Free survival at 12 months | 12 months
Toxicities and feasibility | 15 Weeks
  To assess toxicities and feasibility in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vergnengre, MD, Study Chair — University Hospital, Limoges
Locations (30):
- France (30):
  - Service de Pneumologie, CHU Angers, Angers
  - Service de pneumologie; Centre Hospitalier d'Annecy, Annecy
  - Service de Pneumologie; Centre Hospitalier, Beauvais
  - Service de Pneumologie, Beauvais
  - Service de Pneumologie, Bordeaux
  - CHU Brest, Brest
  - Service de Pneumologie, Charleville Mezière
  - Service de Pneumologie ; Centre hospitalier, Charleville-Mézières
  - Service de Pneumologie, Créteil
  - Service de Pneumologie; Centre Hospitalier, Draguignan
  - Service de Pneumologie, Draguignan
  - Service de Pneumologie, Elbeuf
  - Service de Pneumologie, Gap
  - Département de Pathologie Respiratoire du CHU de Limoges, Limoges
  - Service de Pneumologie, Hôpital de la Croix Rousse, Lyon
  - Service de Pneumologie-Neurologie ; Centre Hospitalier F. Quesnay, Mantes-la-Jolie
  - Département des Maladies Respiratoires ; Hôpital Sainte Marguerite, Marseille
  - CH de Meaux, Meaux
  - Service de Pneumologie, Meaux
  - Service de Pneumologie, Mulhouse
  - Service de Pneumologie - Hôpital St Antoine, Paris, Paris
  - Service de Pneumologie-Allergologie; Centre Hospitalier Général, Périgueux
  - CHU Reims, Reims
  - Service de Pneumologie, Hôpital Pontchailloux, Rennes
  - Service de Pneumologie; CHG de Roanne, Roanne
  - Clinique Pneumologique; Hôpital Charles Nicolle, Rouen
  - Service de Pneumologie; Hôpital Bois Guillaume, Rouen
  - Hôpital Charles Nicolle, Service de Pneumologie, Rouen
  - Service de Pneumologie, Hôpital Nord, Saint-Etienne
  - Service de Pneumologie, Villefranche